CLINICAL TRIAL: NCT04463563
Title: Cerebral Oximetry in Adult Cardiac Surgery to Reduce the Incidence of Neurological Impairment and Hospital Length-of-stay: A Prospective, Randomized, Controlled Trial
Brief Title: Cerebral Oximetry in Cardiac Surgery to Reduce Neurological Impairment and Hospital Length-of-stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: The Hull and East Riding Cardiac Trust Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC-10/H0906/72
Record Dates: First submitted 2020-06-20; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Surgery; Neural Injury; Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Intervention Model Description: This prospective, single centre, double-blinded controlled study randomized 182 consecutive patients, scheduled for cardiac surgical procedures using cardiopulmonary bypass. Participants were randomized by concealed envelope.
Who Masked: Participant, Outcomes Assessor
Masking Description: The personnel assessing and collecting the post-operative data were unaware of the patient group in the operating room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NIRS group. Brain oxygen saturations group. (Active Comparator): A monitor by means of non-invasive stickers will display cerebral oximetry (brain oxygen saturations) throughout the heart surgery.This gives a direct reading of brain frontal lobe oxygen levels. The baseline is recorded before the patient goes to sleep (anaesthetised) and throughout the surgery and time on cardiopulmonary bypass if the brain oxygen levels fall below baseline then various physiological changes are made to restore oxygen to baseline.
  Interventions: Other: Physiological
- Standard Patient Monitoring (No Intervention): No cerebral monitoring. Standard patient monitoring according to normal practice at Castle Hill Hospital apply.

INTERVENTIONS:
Other: Physiological — Changes to carbon dioxide, oxygen flow, cardiac output, blood pressure, haemoglobin, surgical surveillance, depth of anaesthesia, patient position.
  Arms: NIRS group. Brain oxygen saturations group.

SUMMARY:
Cerebral oximetry using near-infrared spectroscopy (NIRS) has been shown to reduce the incidence of neurological dysfunction and hospital length-of-stay in adult cardiac surgery though not all studies agree. A previous audit using cerebral saturations at or above baseline showed improved neurological and length-of-stay outcomes.

DETAILED DESCRIPTION:
This prospective, single centre, double-blinded controlled study randomized 182 consecutive patients, scheduled for cardiac surgical procedures using cardiopulmonary bypass. Participants were randomized by concealed envelope prior to anaesthesia. NIRS study group were managed perioperatively using our NIRS protocol. The control group had standard management without NIRS. Primary outcomes were post-operative neurological impairment and hospital length-of-stay. Secondary outcomes included ventilation times, intensive care unit length-of-stay, major organ dysfunction and mortality

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective cardiac surgery using cardiopulmonary bypass. Patient over 18 years age. -

Exclusion Criteria:

Emergency surgery. Cardiac surgery without cardiopulmonary bypass. Inability to perform test.

Persistent neurological conditions:

Recent stroke. Dementia. Alzheimer's Disease Parkinson's Disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Hospital length-of-stay | Measured in days from the day of operation to the day the patient is discharged from hospital or death in hospital. If neither has occurred within 6 months of participant's operation it will be recorded as 6 months hospital stay.
  How long before discharge post-operatively.
Physical neurological examination | 3 day post-operatively
  Mobility and conscious control of limbs.
Neurological assessment. | 6 months post-operatively
  Telephone interview to assess patients perception of mobility, function and well being. (see below details)
Neurocognitive test 1 | Day 3 post op.
  Fluency and cognitive functions: Mini-Mental State Examination (MMSE). This test is conducted as a questionnaire of 11 questions. Questions include 'what is the date?', 'name the town you are in?', spelling-forwards and backwards, counting backwards, copying a picture, follow an instruction, naming objects etc. The test is scored out of 30 and recorded in a table. The test is repeated on the third post op day and the 2 scores compared to give a number which relates to performance.
Neurocognitive Test 2 | Day 3 post op
  Visual attention and task switching: Trail Making test A and B
Neurocognitive test 3 | Day 3 post op
  Visual-spatial, frontal lobe: Anti-saccadic eye test
Neurocognitive test 4 | Day 3 post op
  Executive function/verbal immediate and delayed recall: Hopkins Verbal and Hopkins Delay.
Neurocognitive test 5 | Day 3 post op
  General well-being HADS (hospital anxiety and depression score) A and D. HADS A -hospital anxiety and depression score relating to Anxiety. HADS D- hospital anxiety and depression score relating to Depression. Patients are asked a question and their response is scored from 0-3. There are 14 questions the score is recorded and compared with the score after the same questions on the 3rd post-op day. The result gives an indication of the patient's mental state and how it may have changed dur to the sugery.
Late neurocognitive test 1.Telephone questionnaire using elements of the previously used questionnaires. | 6 months post op
  General health questions were: how is your overall health, memory, mood, motor function?Designed to be shorter and not require any visual skills. The questions include the patients perception of whether they believe in each domain that their performance is the same, better or worse than before the surgery.
Late neurocognitive test 2. Telephone questionnaire using elements of the previously used questionnaires. | 6 months post op
  Cognition questions were: Date, repeat and recall, serial 7s, spell, recall. Designed to be shorter and not require any visual skills. The questions include the patients perception of whether they believe in each domain that their performance is the same, better or worse than before the surgery.
Late neurocognitive test 3 | 6 months post op
  Functionality questions were: Stairs, driving, cleaning, dressing, eating/cooking.

SECONDARY OUTCOMES:
Intensive Care length-of-stay | The assessment period is every day on ICU until participant moved to ward. Or patient dies on ICU. Total assessment period 6 months.
  Days on ICU. The time from the day of surgery to the discharge to the ward or death. assessed .
Major organ dysfunction | Before hospital discharge
  Renal function is assessed measuring creatinine. Gastrointestinal function is assessed by the diagnosis of ileus or ischaemic bowel at laparotomy. Cardiac function is assessed by the requirement for inotropic support. Respiratory function is assessed by the requirement for ventilation. All these outcomes are have clinical relevance during the stay on ICU.
Mortality | Day of surgery to death. If the participant is discharged from hospital alive it is not a mortality. Assessed for 6 months from the day of surgery.
  Death in hospital at any time following surgery. Death is considered a mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Sean R Bennett, MB Chb, Principal Investigator — Consultant Anaesthetist Hull Hospital Trust

IPD SHARING:
Plan to Share IPD: No